CLINICAL TRIAL: NCT06214858
Title: To Evaluate the Safety, Tolerability, Pharmacokinetics and Food Effects of SHEN211 Tablet in Healthy Subjects With Fasting Single or Multiple Oral Administration
Brief Title: The Safety, Tolerability, Pharmacokinetics and Food Effects of SHEN211 Tablet in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: JKT Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEU-1001
Record Dates: First submitted 2023-12-12; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-12

CONDITIONS: Phase 1
Keywords: SHEN211; Safety; tolerability; pharmacokinetics; food effects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- （Trial group）-SHEN211 tablets (Experimental): part 1：Four dose groups were set up: 110mg,330mg, 550mg and 770mg, each group was intended to include 2 subjects and was administered orally. SHEN211 tablets in the corresponding dose group were given on fasting in the morning of D1. PK blood collection and related tests were completed on day 8 (D8), PK and safety tests were completed on day 10 (D10), and telephone follow-up was performed on day 14 (D14±1).
  part 2：Two dose groups were set up with 8 subjects in each group. In the first dose group, 330mg SHEN211 tablets D1 and 110mgSHEN211 tablets D2 ~ D5 were taken orally once a day (QD). The second dose group was taken orally 660mg SHEN211 tablets on D1 and 220mg SHEN211 tablets from D2 to D5, once a day (QD). PK samples were collected before and after administration, and safety observation was performed up to 8 days after the last administration.
  Interventions: Drug: SHEN211 tablets
- （Placebo group）-placebo tablets (Placebo Comparator): part 1：Four dose groups were set up: 110mg,330mg, 550mg and 770mg, each group was intended to include 2 subjects and was administered orally. placebo tablets in the corresponding dose group were given on fasting in the morning of D1. PK blood collection and related tests were completed on day 8 (D8), PK and safety tests were completed on day 10 (D10), and telephone follow-up was performed on day 14 (D14±1).
  part 2：Two dose groups were set up with 8 subjects in each group. In the first dose group, 330mg placebo tablets D1 and 110mg placebo tablets D2 ~ D5 were taken orally once a day (QD). The second dose group was taken orally 660mg placebo tablets on D1 and 220mg placebo tablets from D2 to D5, once a day (QD). PK samples were collected before and after administration, and safety observation was performed up to 8 days after the last administration.
  Interventions: Drug: SHEN211 placebo tablets
- （Food influence group）-SHEN211 tablets (Experimental): The dose of SHEN211 tablets 330mg was intended to be selected in this experiment. Subjects in group A took SHEN211 tablets 330mg orally on an empty stomach in the morning of the first day of the experiment (the first cycle). On the morning of the 12th day of the trial (the second cycle), SHEN211 tablets 330mg were taken orally once, 30min after starting to eat a high-fat high-calorie meal; Subjects in group B took SHEN211 tablets 330mg orally once in the morning of the first day of the trial (the first cycle) when they started to eat A high-fat and high-calorie meal for 30min, and took SHEN211 tablets 330mg orally in the morning of the 12th day of the trial (the second cycle) on an empty stomach.
  Interventions: Drug: SHEN211 tablets

INTERVENTIONS:
Drug: SHEN211 tablets — SHEN211 tablets, tablets, specification: 0.11g, 10 tablets/box, storage: sealed, not more than 25℃ storage.
  Arms: （Food influence group）-SHEN211 tablets; （Trial group）-SHEN211 tablets
Drug: SHEN211 placebo tablets — placebo tablets, tablets, specification: 0g, 10 tablets/box, storage: sealed, not more than 25℃ storage.
  Arms: （Placebo group）-placebo tablets

SUMMARY:
This is a study to evaluate the safety, tolerability, pharmacokinetics, and food effects of SHEN211 tablet in healthy subjects after fasting single or multiple oral administration

DETAILED DESCRIPTION:
The whole trial consisted of three parts: Part 1 was a single-center, randomized, double-blind, placebo-controlled, single-dose dose increasing safety, tolerability and pharmacokinetic test; Part 2 was a single-center, randomized, double-blind, placebo-controlled, multiple-dose safety, tolerability and pharmacokinetic study. Part 3 is a single-dose, randomized, open, two-phase, double-cross, two-sequence design trial of the effects of food on the main PK parameters of SHEN211 tablets in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy subjects, ages 18-55 (including boundary values)
* The body weight of male subject is not less than 50.0kg, the body weight of female subject is not less than 45.0kg,Body mass index(BMI) in the range of 19.0 ~28.0kg/m2[BMI= weight (kg)/height 2 (m2)] (including the critical value)
* Subjects (including male subjects) are willing to be childfree from screening until 6 months after the last dose of the study drug, voluntarily use effective contraception (see Appendix I), and have no sperm donation plans; Women of childbearing age had to be assessed by a specialist as not pregnant and within 7 days of the start of their last menstrual period before enrollment.
* Sign informed consent before screening, fully understand the test content, process and possible adverse reactions, and be able to complete the study according to the requirements of the test protocol.

Exclusion Criteria:

* Vital signs examination, physical examination, clinical laboratory examination (blood routine, urine routine, blood biochemistry), coagulation function, infection marker examination, pregnancy examination (female only),12-lead electrocardiogram examination, chest X-ray examination, were determined by the investigator to be abnormal and clinically significant
* Any medical history or present medical history that may affect the subject's safety evaluation or study of the drug in vivo process, including but not limited to neurological/psychiatric, respiratory, cardiovascular and cerebrovascular systems, digestive system (any history of gastrointestinal disorders that affect drug absorption), blood and lymphatic system, liver and kidney function, endocrine system, and immune system disorders
* Those who had surgery within 3 months prior to screening or planned to have surgery during the study period, and those who had surgery that would affect drug absorption, distribution, metabolism, or excretion;
* Have a history of allergies to food, drugs, etc., or are known to be allergic to any component of this product
* People who have used any prescription drugs, over-the-counter drugs, Chinese herbs and health products within 2 weeks before screening;
* Any drug that inhibits or induces liver metabolism of drugs (e.g., inducers - barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole) used within 28 days prior to screening; Inhibitors -SSRI antidepressants, cimetidine, Diltiazem, macrolides, nitroimidazoles, sedatives and hypnotics, verapamil, fluoroquinolones, antihistamines);
* Those who received vaccination within 1 month prior to screening or planned to receive vaccination during the study period;
* Those who consumed an average of more than 14 units of alcohol per week (1 unit of alcohol ≈360mL beer or 45mL spirits with 40% alcohol or 150mL wine) in the three months prior to screening, or could not abstain during the test period, or had a positive alcohol breath at baseline;
* People who smoked an average of more than 5 cigarettes per day in the 3 months prior to the first administration of the study drug, or who could not stop using any tobacco products during the trial period;
* Blood donation or blood loss (≥400mL) within 3 months before screening, or blood transfusion;
* Those with a history of drug abuse within 6 months prior to screening;
* Those who had used drugs in the 3 months prior to screening, or who had positive urine screening at baseline;
* Participated in other drug clinical trials within 3 months prior to screening;
* Excessive daily consumption of tea, coffee and/or caffeinated beverages (more than 8 cups on average, 1 cup ≈250mL) in the 3 months before screening;
* Those who have special dietary requirements and cannot accept a unified diet;
* Dysphagia;
* Those with a history of infection (except a history of infection with the novel coronavirus);
* People who are lactose intolerant (those who have had diarrhea from drinking milk);
* Patients who cannot tolerate venipunction or have a history of needle fainting or blood fainting;
* Female subjects who are pregnant or breastfeeding;
* Participants considered inappropriate for clinical trials.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-04-02 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to day 63
  Safety and Tolerability as assessed by AEs and SAEs

SECONDARY OUTCOMES:
Tmax | Up to day 63
  Peak time: The time required to reach peak concentration after administration
Cmax | Up to day 63
  Peak concentration: The highest blood concentration after administration
AUC | Up to day 63
  Area under the drug time curve: The area surrounded by the blood concentration curve to the time axis.
λz | Up to day 63
  Terminal elimination rate: The terminal elimination rate constant is obtained from the semilog linear regression of the phase elimination concentration point
t1/2 | Up to day 63
  Terminal elimination half-life: The time required for the terminal phase blood concentration to decrease by half

CONTACTS AND LOCATIONS:
Overall Officials: wei zhao, ph.D, Principal Investigator — University of Paris 5 - Rene Descartes
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital, Shandong Province), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No